CLINICAL TRIAL: NCT04627675
Title: CORVax12 - a Phase I Trial of SARS-CoV-2 Spike (S) Protein Plasmid DNA Vaccine (CORVax) +/- pIL-12 (Tavokinogene Telseplasmid) in Healthy Volunteers, With Immunodynamic Biomarker Monitoring of Coordinated Cellular/Humoral Response
Brief Title: CORVax12: SARS-CoV-2 Spike (S) Protein Plasmid DNA Vaccine Trial for COVID-19 (SARS-CoV-2)
Acronym: CORVax12
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was ended prematurely due to lack of efficacy. As per FDA guidance, our site continued to follow enrolled subjects through the 180 day safety visit.
Sponsor: Providence Health & Services (Other)
Collaborators: OncoSec Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020000320 CORVax12
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- 1A: Age 18-50; CORVax (Experimental): Healthy volunteers age 18-50 will receive CORVax
  Interventions: Drug: CORVax; Device: Cliniporator
- 1B: Age 18-50; CORVax + pIL-12 (Experimental): Healthy volunteers age 18-50 will receive CORVax + pIL-12
  Interventions: Drug: CORVax; Drug: IL-12 plasmid; Device: Cliniporator
- 2A: Age > 50; CORVax (Experimental): Healthy volunteers age > 50 will receive CORVax
  Interventions: Drug: CORVax; Device: Cliniporator
- 2B: Age > 50; CORVax + pIL-12 (Experimental): Healthy volunteers age > 50 will receive CORVax + pIL-12
  Interventions: Drug: CORVax; Drug: IL-12 plasmid; Device: Cliniporator

INTERVENTIONS:
Drug: CORVax — DNA-encodable coronaviral vaccine
Drug: IL-12 plasmid — cytokine
  Arms: 1B: Age 18-50; CORVax + pIL-12; 2B: Age > 50; CORVax + pIL-12
Device: Cliniporator — electroporation system

SUMMARY:
This is a Phase 1, open-label study to evaluate the safety profile of CORVax +/- pIL-12, (electroporated SARS-CoV-2 spike (S) protein plasmid DNA vaccine with or without the combination of electroporated IL-12p70 plasmid.

DETAILED DESCRIPTION:
This is a Phase 1, open-label study to evaluate the safety profile of CORVax +/- pIL-12, (electroporated SARS-CoV-2 spike (S) protein plasmid DNA vaccine with or without the combination of electroporated IL-12p70 plasmid), given as prime & boost doses, four weeks apart, in healthy volunteers, divided into age groups of 18-50 versus > 50 years old. IL-12p70 plasmid DNA electroporation (tavokinogene telseplasmid) has been extensively studied in over 209 subjects across 11 trials including later stage human cancer trials with more than 1000 administrations. The IGEA CLINIPORATOR® system is approved for clinical use in Europe, but remains investigational in this study.

One participant will initially be enrolled to each of four cohorts and monitored over a 7-day DLT window:

1A. Age 18-50; CORVax.

1. B. Age 18-50; CORVax + pIL-12.
2. A. Age > 50; CORVax.

2B. Age > 50; CORVax + pIL-12.

If after 7 days, no DLT are observed, the cohort may proceed to enroll a second participant. If after monitoring the second participant for 7 days, no DLT are observed, the cohort may proceed to enroll a third participant. If after monitoring the third participant for 7 days, no DLT are observed, the cohort may proceed to enroll six additional participants, for a total of nine participants per cohort using a (1+1+1, +6) design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers ages 18 years and above, who are able to provide written informed consent and willing to allow storage and future use of samples for SARS-CoV-2 related research.
* Women of childbearing potential (WOCBP) must have negative serum or urine pregnancy on each day of vaccine administration.
* Males and women of childbearing potential must agree to take appropriate precautions to avoid pregnancy during treatment and through 180 days after last dose of IP.

Exclusion Criteria:

* Current or previous SARS-CoV-2 infection or receipt of an experimental treatment for prevention of SARS-CoV-2.
* Administration of any vaccine within 4 weeks of first dose.
* Any laboratory abnormalities at baseline greater than Grade 1 per the "FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials": https://www.fda.gov/regulatory-information/search-fda-guidance-documents/toxicity-grading-scale-healthy-adult-and-adolescent-volunteers-enrolled-preventive-vaccine-clinical
* Any history of cardiac arrhythmia.
* Any history of epilepsy or seizure within the last five years.
* Use of immunosuppressive medication within 14 days before the first dose of study drug.
* Anticipated treatment with TNF-α inhibitors (e.g., infliximab, adalimumab, or etanercept).
* Pregnancy or breastfeeding.
* Body mass index of 35 kg/m2 or more.
* Administration of any monoclonal or polyclonal antibody product within 4 weeks of the first dose.
* Chronic liver disease or cirrhosis.
* Previous major surgery or any radiation therapy within 4 weeks of group assignment.
* Any pre-excitation syndromes (e.g., Wolff- Parkinson-White syndrome).
* Metal implants within 20cm of the planned site(s) of injection; presence of keloid scar formation or hypertrophic scar as a clinically significant medical condition at the planned site(s) of injection; tattoos covering the injection site area.
* Presence of a cardiac pacemaker or automatic implantable cardioverter defibrillator.
* History of allogeneic organ transplantation.
* History of primary immunodeficiency.
* Known HIV, hepatitis B virus, or hepatitis C virus infection. Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.
* Uncontrolled intercurrent illness, including but not limited to symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, unstable cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the participant to give written informed consent.
* Comorbidities, controlled or otherwise, associated with higher risk for severe COVID-19 illness - because our understanding of the pathogenesis of SARS-CoV-2 continues to evolve, this will be based on most current information available at time of screening regarding risk factors for severe disease, using resources such as those described on the Centers for Disease Control website: https://www.cdc.gov/coronavirus/2019-ncov/need-extra-precautions/people-at-higher-risk.html
* Subjects at high-risk for SARS-CoV-2 exposure per investigator, including healthcare workers, first responders, and individuals with known exposure to individuals infected with SARS-CoV-2.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice).
* History of autoimmune or inflammatory disorders including but not limited to inflammatory bowel disease (e.g., colitis or Crohn's disease), diverticulitis (with the exception of diverticulosis), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, (see Appendix 2).
* Known allergy or hypersensitivity to study drug(s) or compounds of similar biologic composition to the study drug(s), or any of the study drug excipients.
* Investigator discretion relating to any condition which might interfere with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated prematurely due to lack of efficacy. Per FDA guidance, enrolled patients were followed until Day 180 for safety.
Period: Overall Study
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Started | 3 | 3 | 2 | 3
Completed | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 16 patients were enrolled into the study, however 1 withdrew prior to treatment and 4 were found ineligible during the screening visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12 | Total
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 3 | 11
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 1 | 4
  Male | 1 | 2 | 2 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 2 | 9
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 2 | 1 | 8
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 2 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Occurring on Day 1
Description: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (Grade 1 mild is the minimum value and Grade 4 life threatening is the maximum value.)
Time Frame: Day 1
Population: Study was terminated prematurely due to lack of efficacy. Per FDA guidance, enrolled patients were followed until Day 180 for safety.
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants
  Grade 1 | 2 | 1 | 0 | 1
  Grade 2 | 0 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events Occurring on Day 2
Description: as for outcome 1
Time Frame: Day 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants
  Grade 1 | 1 | 3 | 0 | 1
  Grade 2 | 0 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Adverse Events Occurring on Day 3
Description: as for outcome 1
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants
  Grade 1 | 1 | 1 | 0 | 0
  Grade 2 | 1 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Adverse Events Occurring on Day 15
Description: as for outcome 1
Time Frame: Day 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants
  Grade 1 | 2 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 1
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Adverse Events Occurring on Day 30
Description: as for outcome 1
Time Frame: Day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants
  Grade 1 | 1 | 2 | 1 | 1
  Grade 2 | 0 | 2 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Adverse Events Occurring on Day 31
Description: as for outcome 1
Time Frame: Day 31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants
  Grade 1 | 0 | 2 | 2 | 0
  Grade 2 | 0 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Adverse Events Occurring on Day 32
Description: as for outcome 1
Time Frame: Day 32
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants
  Grade 1 | 1 | 2 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Adverse Events Occurring on Day 45
Description: as for outcome 1
Time Frame: Day 45
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants
  Grade 1 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Adverse Events Occurring on Day 60
Description: as for outcome 1
Time Frame: Day 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants
  Grade 1 | 0 | 1 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Adverse Events Occurring on Day 90
Description: as for outcome 1
Time Frame: Day 90
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants
  Grade 1 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

11. Primary Outcome: Medically Attended Adverse Events (MAAEs)
Description: Extended monitoring of Medically Attended Adverse Events (MAAEs) for potentially immune-mediated conditions (pIMMCs).
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants | 0 | 0 | 0 | 0

12. Primary Outcome: Medically Attended Adverse Events (MAAEs)
Description: Extended monitoring of Medically Attended Adverse Events (MAAEs) for potentially immune-mediated conditions (pIMMCs)
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants | 0 | 0 | 0 | 0

13. Primary Outcome: Medically Attended Adverse Events (MAAEs)
Description: Extended monitoring of Medically Attended Adverse Events (MAAEs) for potentially immune-mediated conditions (pIMMCs)
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants | 0 | 0 | 0 | 0

14. Primary Outcome: Medically Attended Adverse Events (MAAEs)
Description: Extended monitoring of Medically Attended Adverse Events (MAAEs) for potentially immune-mediated conditions (pIMMCs)
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants | 0 | 0 | 0 | 0

15. Primary Outcome: Medically Attended Adverse Events (MAAEs)
Description: Extended monitoring of Medically Attended Adverse Events (MAAEs) for potentially immune-mediated conditions (pIMMCs)
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants | 0 | 0 | 0 | 0

16. Primary Outcome: Medically Attended Adverse Events (MAAEs)
Description: Extended monitoring of Medically Attended Adverse Events (MAAEs) for potentially immune-mediated conditions (pIMMCs)
Time Frame: Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For adverse events, up to Day 90. For medically attended adverse events, starting at Day 30 to Month 18.
Arm/Group | 1A: Age 18-50; CORVax | 1B: Age 18-50; CORVax + pIL-12 | 2A: Age > 50; CORVax | 2B: Age > 50; CORVax + pIL-12
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1A: Age 18-50; CORVax (N=3) | 1B: Age 18-50; CORVax + pIL-12 (N=3) | 2A: Age > 50; CORVax (N=2) | 2B: Age > 50; CORVax + pIL-12 (N=3)
Increased CPK (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1A: Age 18-50; CORVax (N=3) | 1B: Age 18-50; CORVax + pIL-12 (N=3) | 2A: Age > 50; CORVax (N=2) | 2B: Age > 50; CORVax + pIL-12 (N=3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased hemoglobin (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Elevated creatinine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 2 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased BUN (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased CPK (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site redness (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain at electroporation site (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Pain at injection site (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Pruritus at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reduced appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT04627675/Prot_SAP_000.pdf